CLINICAL TRIAL: NCT01496079
Title: The Role of Immunizing Pregnant Women In Protecting Young Infants Against Influenza
Brief Title: Maternal Immunization: Giving Immunity For Tomorrow
Acronym: MI GIFT
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Julie Shakib, Assistant Professor of Pediatrics, Principal Investigator, University of Utah
Other Study IDs: 00051718
Record Dates: First submitted 2011-11-28; First posted 2011-12-21 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Pregnancy; Influenza
Keywords: Maternal immunization; Infant immunization; Influenza vaccine; Passive transfer of immunity
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Inactivated influenza vaccine in pregnancy: Healthy pregnant women who elect to receive inactivated influenza vaccine in early pregnancy (< 20 weeks gestation) and their infants
- No inactivated influenza vaccine during pregnancy: Healthy pregnant women who decline inactivated influenza vaccine in pregnancy and their infants

SUMMARY:
Study objectives are to compare

* influenza antibody levels in infant sera and maternal colostrum or breast milk at delivery, 2, and 6 months women who receive influenza immunization in early pregnancy, late pregnancy, or no influenza immunization during pregnancy and their infants

Study hypotheses are that infants born to pregnant women who receive influenza immunization in late pregnancy will have

* higher levels and a longer serum influenza antibody duration in sera (hemagglutination inhibition (HAI) titers) and colostrum/breast milk (influenza-specific IgA and IgG by enzyme-linked immunosorbent assay (ELISA) than infants of women immunized in early pregnancy or not immunized

ELIGIBILITY:
Inclusion Criteria:

Pregnant women 18-45 years of age from 8-36 weeks gestation in good health as determined by medical history and recent physical exam who

* receive prenatal care at the UUHS Obstetrics and Gynecology Clinics and their infants
* plan to seek care for their infant at the UUHS affiliated Pediatric Clinics (UUHS or SMC Pediatric Clinics)
* plan for their infant to receive influenza immunization at 6 and 7 months of age

Exclusion Criteria:

* maternal history of either a congenital or acquired immunodeficiency including infection (e.g. HIV), chronic steroid use, or malignancy
* serious underlying neurological, cardiac, renal, or pulmonary disease in either the mother or infant
* multiple gestation
* antenatal or postnatal detection at delivery of any major birth defect in the infant
* delivery of the infant before 37 weeks

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women and their infants receiving care at University of Utah Health Sciences (UUHS) will be recruited and followed.
Sampling Method: Non-Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2011-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Influenza antibody titer levels in infants born to women who receive inactivated influenza vaccine in early pregnancy compared with late pregnancy and no immunization | Infant antibody titers at delivery
  Influenza titers will be measured on infant serum and breast milk samples by HAI assay and on maternal colostrum or breast milk if available by ELISA and neutralization assay

CONTACTS AND LOCATIONS:
Overall Officials: Julie H. Shakib, DO, MS, MPH, Principal Investigator — University of Utah
Locations (1):
- University of Utah Health Sciences Center, Salt Lake City, Utah, United States